CLINICAL TRIAL: NCT01495013
Title: Study ATG115317, a Comparison of Atorvastatin and Glimepiride Fixed Dose Combination and Atorvastatin and Glimepiride Loose Combination in the Treatment of Patients With Type 2 Diabetes Mellitus
Brief Title: A Comparison of Atorvastatin and Glimepiride Fixed Dose Combination and Atorvastatin and Glimepiride Loose Combination in the Treatment of Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115317
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: non-inferiority; glimepiride; LDL cholesterol; fixed dose combination; atorvastatin; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — glimepiride; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glimepiride Atorvastatin fixed dose combination (Active Comparator): All subjects will start on 1mg glimepiride/10 mg atorvastatin fixed dose combination (FDC) and either treatment can be titrated up based on fasting glucose or LDL levels. The following glimepiride/atorvastations FDCs will be available for use 1mg/10mg, 2mg/10mg, 3mg/10mg, 4mg/10mg, 1mg/20mg, 2mg/20mg, 3mg/20mg, 4mg/20mg.
  Interventions: Drug: 1mg Glimepiride/10mg Atorvastatin FDC; Drug: 2mg Glimepiride/10mg Atorvastatin FDC; Drug: 3mg Glimepiride/10mg Atorvastatin FDC; Drug: 4mg Glimepiride/10mg Atorvastatin FDC; Drug: 1mg Glimepiride/20mg Atorvastatin FDC; Drug: 2mg Glimepiride/20mg Atorvastatin FDC; Drug: 3mg Glimepiride/20mg Atorvastatin FDC; Drug: 4mg Glimepiride/20mg Atorvastatin FDC
- Glimepiride +Atrovastatin loose combination (Active Comparator): All subjects will start on 1mg glimepiride/10 mg atorvastatin loose combination (given as separate tablets) and either treatment can be titrated up based on fasting glucose or LDL levels. Glimepiride single dose tablets are available for 1mg, 2mg, 3mg and 4mg. Atorvastatin single dose tablets are available for 10mg and 20mg.
  Interventions: Drug: 1mg Glimepiride; Drug: 2mg Glimepiride; Drug: 3mg Glimepiride; Drug: 4mg Glimepiride; Drug: 10mg Atorvastatin; Drug: 20mg Atorvastatin

INTERVENTIONS:
Drug: 1mg Glimepiride/10mg Atorvastatin FDC — 1 tablet by mouth once a day
  Arms: Glimepiride Atorvastatin fixed dose combination
Drug: 2mg Glimepiride/10mg Atorvastatin FDC — 1 tablet by mouth once a day
  Arms: Glimepiride Atorvastatin fixed dose combination
Drug: 3mg Glimepiride/10mg Atorvastatin FDC — 1 tablet by mouth once a day
  Arms: Glimepiride Atorvastatin fixed dose combination
Drug: 4mg Glimepiride/10mg Atorvastatin FDC — 1 tablet by mouth once a day
  Arms: Glimepiride Atorvastatin fixed dose combination
Drug: 1mg Glimepiride/20mg Atorvastatin FDC — 1 tablet by mouth once a day
  Arms: Glimepiride Atorvastatin fixed dose combination
Drug: 2mg Glimepiride/20mg Atorvastatin FDC — 1 tablet by mouth once a day
  Arms: Glimepiride Atorvastatin fixed dose combination
Drug: 3mg Glimepiride/20mg Atorvastatin FDC — 1 tablet by mouth once a day
  Arms: Glimepiride Atorvastatin fixed dose combination
Drug: 4mg Glimepiride/20mg Atorvastatin FDC — 1 tablet by mouth once a day
  Arms: Glimepiride Atorvastatin fixed dose combination
Drug: 1mg Glimepiride — 1 tablet of Glimepiride and 1 tablet of Atorvastatin co-administered once daily
  Arms: Glimepiride +Atrovastatin loose combination
Drug: 2mg Glimepiride — 1 tablet of Glimepiride and 1 tablet of Atorvastatin co-administered once daily
  Arms: Glimepiride +Atrovastatin loose combination
Drug: 3mg Glimepiride — 1 tablet of Glimepiride and 1 tablet of Atorvastatin co-administered once daily
  Arms: Glimepiride +Atrovastatin loose combination
Drug: 4mg Glimepiride — 1 tablet of Glimepiride and 1 tablet of Atorvastatin co-administered once daily
  Arms: Glimepiride +Atrovastatin loose combination
Drug: 10mg Atorvastatin — 1 tablet of Atorvastatin and 1 tablet of Glimepiride co-administered once daily
  Arms: Glimepiride +Atrovastatin loose combination
Drug: 20mg Atorvastatin — 1 tablet of Atorvastatin and 1 tablet of Glimepiride co-administered once daily
  Arms: Glimepiride +Atrovastatin loose combination

SUMMARY:
The aim of this 20 week study is to show that glimepiride/atorvastatin fixed dose combination tablet is safe and as effective as atorvastatin + glimepiride combination taken as separate tablets, in improving glycaemic control (glycated haemoglobin, HbA1c) and cholesterol levels (Low-density lipoprotein, LDL) in diabetic subjects, who are inadequately controlled on a stable dose of metformin. Eight dose combinations will be included.

DETAILED DESCRIPTION:
Patients diagnosed with Type 2 diabetes (T2D) are initially provided with lifestyle advice in order to manage the condition by diet, exercise and weight reduction, followed by treatment with metformin. However, many patients do not gain adequate control of fasting glucose by these methods and other anti-diabetic agents are needed. Furthermore, these patients have an increased cardiovascular risk compared with the general population. Approximately one half of patients with T2D die prematurely of a cardiovascular cause and approximately 10% die of renal failure.

Atherogenic dyslipidemia, which is defined as the triad of elevated triglycerides, low high-density lipoprotein cholesterol (HDL-C), and small low-density lipoprotein cholesterol (LDL-C) particles, is commonly found in individuals with T2D. In diabetic patients, the LDL particles tend to be smaller, denser, and more atherogenic than in the general population. As a result, in patients with diabetes, lowering LDL-C levels may lead to a greater benefit in terms of Cardiovascular disease (CVD) risk reduction than in patients without diabetes. Multiple clinical trials have demonstrated significant benefits of lipid-lowering (primarily statin) therapy on CVD outcomes for primary and secondary prevention, irrespective of baseline lipid levels. Hence, clinical treatment guidelines recommend that patients with T2D should be treated with both an anti-diabetic agent and a statin.

Glimepiride is an established once-daily sulphonylurea for use as first-line therapy, and is often used in patients who are metformin intolerant, or in those who are failing to achieve glucose control on metformin monotherapy. Atorvastatin is an established statin that is indicated for reducing the risk of cardiovascular events in diabetic patients, without clinically evident coronary heart disease (CHD), irrespective of whether cholesterol is raised. The risk:benefit of both glimepiride and atorvastatin is well established and described in the approved product labels. There is widespread use of both glimepiride and atorvastatin, prescribed separately, in the T2D population. The available literature indicates that there is no drug-drug interaction risk associated with this combination therapy and no clinical PK interactions between atorvastatin and glimepiride have been recorded. A once-daily combination product which combines both glimepiride and atorvastatin will fulfil an unmet clinical need in simplifying patient treatment regimens in a patient population who have a significant disease burden. Providing concurrent access to a statin in patients with T2D, in addition to medication to manage glucose levels, is a critical requirement for ensuring appropriate management of cardio-metabolic risk.

In this study, subjects already on a stable dose of metformin will be randomised to either to receive the glimepiride/atorvastatin fixed dose combination treatment or atorvastatin + glimepiride combination taken as separate tablets. The starting dose for all subjects will be 1mg glimepiride and 10mg atorvastatin. The glimepiride dose will be titrated up if the average fasting glucose is >7.0mmol/L. The atorvastatin dose will be titrated up if LDL is >2.6mmol/L.

The purpose of the study is to demonstrate non-inferiority of the glimepiride/atorvastatin fixed dose combination compared with glimepiride +atorvastatin taken as separate tablets in reducing HbA1c and LDL.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) males and females ( including of child-bearing potential) with Type 2 diabetes mellitus.
* Currently treated for Type 2 daibetes mellitus with metformin monotherapy and have been a stable dose of metformin for atleast 3 months
* patients with CVD or ≥40 years old with a cardiovascular risk factor, or <40 years old with LDL-C level 100mg/dL
* HbA1c levels ≥7.0 and <9.5% at screening or within 3 months prior to study enrollment
* Fasting blood glucose >7.0 mmol/L on 4 days in a week
* Statin-naïve or no statin use for 2 months prior to screening
* Provision of informed consent

Exclusion Criteria:

* Concomitant treatment:
* Concomitant treatment with statins other than study medication
* Concomitant treatment with fenofibrate or other lipid lowering agents
* concomitant treatment with anti-diabetic therapy other than study treatment or change in metformin monotherapy for subjects already treated with metformin
* Concurrent diseases and symptoms:
* Subjects with Type 1 diabetes or who have a current need for insulin therapy
* Subjects with symptomatic hyperglycaemia requiring immediate therapy in the judgement of the investigator
* Subjects with myalgia
* Significant hypertriglyceridaemia as defined by fasting triglycerides >3.5 mmol/L
* Clinically significant ongoing cardiovascular disease:
* Subjects who have had an acute cardiovascular event within 30 days prior to randomisation
* Subjects with unstable or severe angina, coronary insufficiency or New York Heart Association class III-IV heart failure
* subjects with a prior heart transplant or who are awaiting a heart transplant
* Subjects with systolic blood pressure >160 mmHg or diastolic blood pressure >90 mmHg while on anti-hypertensive treatment
* General Health:
* Subjects with end stage renal disease requiring renal replacement therapy
* Subjects receiving drug therapy to treat liver disease
* Subjects with diagnosis of cancer ( other than superficial squamous. basal cell skin cancer or adequately treated cervical carcinoma in situ) in the past 3 years or who are currently receiving treatment for an active cancer ( other than prophylactic)
* Subjects with a clinically significant abnormality identified at screening on physical examination or laboratory tests (including thyroid stimulating hormone) which, in the judgement of the investigator, would preclude safe completion of the study
* Subjects with anaemia defined by a haemoglobin concentration <10 g/dL (100) g/L) for females and <12 g/dL (120 g/L) for males or a haemoglobinopathy that could interfere with the assessment of HbA1c
* Subjects with clinically significant liver disease as defined by alanine aminotransferase ( ALT) or aspartate aminotransferase (AST) levels >2.5 times the upper limit of normal (ULN) or a diagnosis of Chronic active hepatitis including that of viral aetiology, or on antiviral or immunosuppressive therapy
* Subjects with contraindications to or history of hypersensitivity to, the investigational products
* Subjects who are clinically or medically unstable, with expected survival <1 year
* Subjects with a recent history ( within the last 6 months ) or suspicion of current drug abuse or alcohol abuse
* Any other factor likely to limit protocol compliance or reporting of adverse events
* Previous study participation:
* Participation in another clinical trial of an investigational agent, if the subject has used an investigational agent within 30 days or 5 half lives (whichever is longer) preceding the Screening Visit
* Previous randomisation in this study

Contraception:

* Females of child-bearing potential who are not using highly effective methods for avoiding pregnancy. Highly effective methods include:
* Oral Contraceptive, either combined or progestogen alone
* Injectable progestogen
* Implants of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches
* Intrauterine device or intrauterine system with a failure rate of less than 1% per year
* Male partner sterilisation (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records
* Double barrier method: condom and an occlusive cap(diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository), including nonoxynol-9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Non inferiority of glimepiride/atorvastatin compared with glimepiride + atorvastatin taken as separate tablets in reducing HbA1c levels | Week 20
  Change from baseline
Non inferiority of glimepiride/atorvastatin compared with glimepiride + atorvastatin taken as separate tablets in reducing LDL levels | Week 20
  Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- Malaysia (4):
  - GSK Investigational Site, Ipoh
  - GSK Investigational Site, Johor Bahru
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kubang Kerian
- Mexico (5):
  - GSK Investigational Site, Cuernavaca
  - GSK Investigational Site, Del. Cuauhtémoc
  - GSK Investigational Site, Gadalajara, Jalisco
  - GSK Investigational Site, Guadalajara Jalisco
  - GSK Investigational Site, Mexico City
- Philippines (5):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Santa Cruz, Manila
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
- South Korea (7):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Kangwondo
  - GSK Investigational Site, Seocho-ku, Seoul
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
- Thailand (3):
  - GSK Investigational Site, Chiangrai
  - GSK Investigational Site, Nakhon Ratchasima
  - GSK Investigational Site, Rajathevee

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 115317 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115317 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115317 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115317 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115317 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115317 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register